CLINICAL TRIAL: NCT00352222
Title: A Prospective, Multicenter, Single Arm Study to Obtain Additional Data on the Safety and Efficacy of the Express Vascular LD Implantation in the Treatment of Stenosed or Occlusive Atherosclerotic Disease in Iliac Arteries
Brief Title: Safety and Efficacy of Express LD to Treat Stenosed or Occlusive Atherosclerotic Disease in Iliac Arteries
Acronym: MELODIE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: KIKA (Unknown)
Responsible Party: Anne Cornaille, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2015; MTE-E-0301
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Arterial Occlusive Disease; Intermittent Claudication; Atherosclerotic Disease; Thrombosis
Keywords: iliac arteries; implantation; treatment of atherosclerotic disease; stenosed; occlusive
MeSH Terms: conditions — Arterial Occlusive Diseases; Intermittent Claudication; Thrombosis; Bites and Stings

INTERVENTIONS:
Device: stent implantation

SUMMARY:
To obtain additional data on safety and efficacy of the Express stent implantation in the treatment of stenosed or occlusive atherosclerotic disease (de novo or restenotic lesions) in the iliac arteries (common or external).

DETAILED DESCRIPTION:
This study was conducted to provide additional data on the safety and efficacy of the Express™ Vascular LD stent, particularly with regard to the long-term patency in iliac arteries. The study would provide data on angiographic endpoints and clinical outcomes at 30 days, 6 months, and at 12 and 24 months post implantation in atherosclerotic lesions in iliac arteries. The data obtained in this study with the use of the Express™ Vascular LD stent was compared with historical data obtained from the use of the Palmaz balloon-expandable stent. The Palmaz balloon expandable stent has been chosen as the control device because it is currently the only FDA-approved balloon-expandable stent for use in the percutaneous treatment of atherosclerotic disease in iliac arteries.

The Palmaz balloon-expandable stent is no longer commercialized in Europe. Therefore a randomized study with the Palmaz balloon-expandable stent was not feasible. In addition, there are no ongoing or published randomized trials describing performance of a newer version of the Palmaz stent in iliac atherosclerotic lesions. In order to adequately compare the efficacy data of the ExpressTM Vascular LD stent with the efficacy data of the Palmaz balloon-expandable stent, the same efficacy parameter as in the publication on the Palmaz balloon-expandable stent was measured in this study: % mean loss of the luminal diameter at 6 months post-procedure.

The findings of the longer-term Follow-Up assessments at 12 and 24 months will be presented as the results from these assessments become available.

ELIGIBILITY:
Inclusion Criteria:

* chronic symptomatic atherosclerotic disease in the iliac arteries (Fontaine Class IIa, IIb, and III)
* atherosclerotic de novo or restenotic lesions in the common and/or external iliac artery.
* baseline diameter stenosis of > or = 50%
* reference vessel diameter > or = 5mm and < or = 10mm
* at least one sufficient ipsilateral infrapopliteal run-off
* length of diseased segment(s) < or = 10cm and can be treated with maximally two overlapping Express Vascular LD Stents.
* multiple target lesions of the iliac arteries in the same patient can be included provided if each target lesion is compliant with the antiographic inclusion criteria and non-compliant with any of the antiographic exclusion criteria, target lesions are not located in the same target axis, and all target lesions can be treated during the same procedure.

Exclusion Criteria:

* chronic symptomatic atherosclerotic disease classified as fontaine Class I or IV
* acute leg ischemia
* pregnants patients
* patients with uncorrected bleeding disorders (platelets < 150 000/mm3 or > 450 000 mm3, or patient who cannot receive anticoagulation or antiplatelet aggregation therapy
* patient with known allergy to stainless steel
* known anaphylactoid or other non-anaphylactic reactions to contrast agents that cannot be adequately premedicated prior to the index procedure
* life-expectancy of less than 24 months due to other medical co-morbid condition that could limit patient's ability to participate in the study, the patient's compliance with the follow-up requirements or impact the scientific integrity of the study
* patient currently participating in another study that has not yet completed the primary endpoint or that clinically interferes with the endpoint of this study
* patients who have already participated in this study
* patients with prior or planned bypass surgery of the target vessel
* patient with prior stent placement in the target vessel
* patient with any previous coronary intervention within the last 30 days before enrollment into this study or patients with planned coronary intervention within 30 days after enrollment into this study.
* patients in whom the origin of the profunda femoris and superficial femoral artery is occluded in the limb supplied by the iliac artery to be treated without planned surgical repair
* patients with heavily calcified and excessive tortuous lesions at the target site as determined by angiography
* patients with target lesion which is within or adjacent to the proximal or distal segment of an aneurysm
* patients with persistent, acute intraluminal thrombus of the proposed target lesion site post-thrombolytic therapy
* patients with perforated vessels as evidenced by extravasation of contrast media
* patients with multiple lesions in the same target vessels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-01; Primary Completion 2005-07 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Angiographic mean percent loss of luminal diameter at 6 months post-procedure defined as ((post-procedure MLD - Follow-up MLD)/Post-procedure MLD) X 100

SECONDARY OUTCOMES:
hemodynamic success at hospital discharge, 30 days and 6, 12 and 24 months post-procedure, angiographic binary restenosis at 6 mont

CONTACTS AND LOCATIONS:
Overall Officials: Luc Stockx, MD, Principal Investigator — Limburgs Vaatcentrum Ziekenhuis Oost-Limburg, Belgium
Locations (10):
- Belgium (2):
  - Limburgs Vaatcentrum Ziekenhuis Oost-Limburg, Genk
  - Sint Trudo Hospital, Sint-Truiden
- CHUM- Notre Dame Hospital, Montreal, Quebec, Canada
- Czechia (2):
  - General Teaching Hospital Prague, Prague
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
- Sint Antonius Hospital, Nieuwegein, CM, Netherlands
- Poland (4):
  - University Hospital of Krakow, Krakow
  - University School of Medicine, Lublin
  - Center of Diagnostic Imaging and Vascular Disease Treatment, Szczecin
  - Samodzielny Publiczny Centraln Szpital, Warsaw

REFERENCES:
- [Derived] Stockx L, Poncyljusz W, Krzanowski M, Schroe H, Allocco DJ, Dawkins KD; MELODIE Investigators. Express LD vascular stent in the treatment of iliac artery lesions: 24-month results from the MELODIE trial. J Endovasc Ther. 2010 Oct;17(5):633-41. doi: 10.1583/09-2917MR.1. PMID 20939723